CLINICAL TRIAL: NCT03996733
Title: The Effectiveness Of Using A Gelatin-Based Model In Ultrasonography Guided Jugular Central Venous Catheter Placement Training
Brief Title: Using A Gelatin-Based Model In USG-Guided Jugular Venous Catheter Placement Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeki Tuncel Tekgul (Other)
Responsible Party: Sponsor-Investigator, Zeki Tuncel Tekgul, Assoc. Prof. Dr, Bozyaka Training and Research Hospital
Organization: Bozyaka Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JugulerUsgMaket
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Central Venous Catheters; Vascular Access Devices; Education; Simulation Training; Ultrasonography, Interventional
Keywords: Training; Education; Homemade; Model; Central Venous Catheterization; Ultrasound Guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GControl (Active Comparator): Participants will attend the lecture for 30 minutes and watch a demo video showing the procedure. Later, they will practice ultrasound imaging of right jugular vein on a real human subject.
  Interventions: Other: Lecture; Other: Demo Video; Other: UltrasoundImaging
- GModel (Experimental): Participants will attend the lecture for 30 minutes and watch a demo video showing the procedure. Later, they will practice ultrasound imaging of right jugular vein on a real human subject.
  Participants in this group will also practice jugular vein puncture on our homemade jugular central venous catheterization training model.
  Interventions: Other: Lecture; Other: Demo Video; Other: UltrasoundImaging; Other: ModelTraining

INTERVENTIONS:
Other: Lecture — Principal investigator of the study will lecture about the ultrasound guided jugular central venous catheterization according to latest guidelines.
Other: Demo Video — Investigators of the study prepared a detailed demo-video showing insertion of a jugular central venous catheter with USG guidance. Principal investigator will vocalize the video in real-time.
Other: UltrasoundImaging — Participants will exercise the proper visualisation of the right jugular vein at T6 level with USG guidance on a human subject.
Other: ModelTraining — Participants will exercise the proper punction of juguler vein with USG guidance on the homemade jugular venous catheterization training model.
  Training model will include carotid artery, trachea and plaure in accordance with the real anatomy.
  Arms: GModel

SUMMARY:
An education model with a homemade jugular venous catheterization model will be compared to the conventional training model for ultrasound-guided central jugular line catheterization.

The study will include 60 residents to be divided into two groups with stratified random sampling.

Training session for the control group (Group 2) will include a lecture about the subject, a demo video presentation, and practice of visualization of right jugular vein on a real human subject.

Training session for the model group (Group 1) will include the same as GControl with the addition of the puncture practice on the homemade jugular venous catheterization model(HJVCM) with ultrasound guidance.

Both groups will be tested with another HJVCM individually and the results of the success and fail parameters will be compared.

DETAILED DESCRIPTION:
According to the latest guidelines, ultrasound guidance has become the golden standard in Jugular Central Venous Catheter applications. This reveals the necessity of theoretical and practical training on USG for jugular central venous catheter training. Models for jugular venous catheterization training are few in number and also expensive. Thus, the investigators built an Homemade Jugular Venous Catheterization Model which meant to be cheap and easy to make and transport. With this study, the investigators will test whether this model will provide any benefit to the success of the training on USG Guided Jugular Venous Catheterization.

Two different training sessions are planned as one will include the training model and the other will not. The study will be conducted with resident physicians without any experience on jugular venous catheterization or ultrasound-guided interventions of any kind. Participants will be divided into two groups with stratified random sampling (According to specialties and years of residency) and the both will attend to a 30 minutes lecture on jugular venous catheterization with US guidance and basic ultrasound principles including a demo video illustrating the procedure. Later, the participants will practice ultrasound imaging of right jugular vein on a real human subject. The model training group will be named Group 1 and control group will be named Group 2. Group 1 will also practice jugular vein puncture on the training model. After training sessions, each participant will be tested with a different model placed in a manikin. The assessment session will include successful visualization of the jugular vein, puncture of the jugular vein, and insertion of the guide wire. Evaluation of the success and fail parameters (explained in outcome parameters) will be monitored by four educated supervisors. The sessions for both of the groups are planned to take 120 minutes in total and the assessment will be limited to five minutes individually.

ELIGIBILITY:
Inclusion Criteria:

* Residents

Exclusion Criteria:

* Any experience on jugular venous catheterization
* Experience of ultrasound guided interventions of any kind.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Success Of The Catheterization | 5 minutes
  Successful visualization of the jugular vein in long axis, successful puncture and draining the fluid in the jugular vein, successful visualization of insertion of the guide wire. All required.

SECONDARY OUTCOMES:
Successful Visualization | 5 minutes
  Successful visualization of the jugular vein in long axis. Yes or No.
Time Of The Successful Visualization | 5 minutes
  Total time from puncture of the model's skin to the successful visualization of the jufular vein in long axis.
Puncture Count | 5 minutes
  Total count of punctures on model skin.
Number Of Changes Of Needle Angle During The Procedure | 5 minutes
  Retraction and orientation of the needle at different angles before the puncture of the jugular vein.
Puncture Time | 5 minutes
  Total time from puncture of the model's skin to the successful puncture of the jugular vein.
Fail Of The Procedure | 5 minutes
  Any of these four endpoints;
  * Puncture of pleura
  * Puncture of carotid artery
  * Puncture of the base(Too deep needle advancement)
  * Exceeding five minutes, before successful jugular venous catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Karabağlar, İzmir, Turkey (Türkiye)